CLINICAL TRIAL: NCT03227536
Title: Asphyxia at Birth : Evolution of Birth Asphyxia Rate, Etiologies and Neonatal Outcome From 2000 to 2016
Brief Title: Asphyxia at Birth : Causes and Neonatal Outcome
Acronym: ABC-NEO
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 17-118
Record Dates: First submitted 2017-07-11; First posted 2017-07-24 (Actual); Last update posted 2017-07-24 (Actual); Status verified 2017-07

CONDITIONS: Neonatal Asphyxia
Keywords: Neonatal asphyxia; neonatal acidosis; fetal ECG; umbilical cord acid-base status
MeSH Terms: conditions — Asphyxia Neonatorum

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is an historic cohort study based on the birth and delivery register of the HFME maternity ward. This study aim at understanding the evolution of asphyxia at birth, at all gestational ages, identifying causes and describing neonatal outcomes since 2000, when a second line strategy for foetal surveillance (fetal ECG) and systematic umbilical acid-gas cord blood were introduced in our maternity ward.

The investigator's hypothesis was that the neonatal asphyxia decrease could be due to 3 main factors including second line strategy introduction, systematic umbilical cord acid-base implementation and improvement in antenatal risk factor screening for asphyxia. The investigator's second hypothesis was that neonatal prognosis in neonates with acidosis was improved with systematic early after birth EEG evaluation, allowing early treatment and surveillance.

ELIGIBILITY:
Inclusion Criteria:

* All births at the maternity ward of the hospital Femme-Mère-Enfant from 1st of january 2000 to 31 december 2016

Exclusion Criteria:

* Infants born after medical pregnancy termination and born out of the hospital and secondarily hospitalized in our department will be excluded

Max Age: 1 Hour | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All births at the maternity ward of the hospital Femme-Mère-Enfant from 1st of january 2000 to 31 december 2016
Sampling Method: Non-Probability Sample
Enrollment: 61448 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Rate of Neonatal asphyxia | 2 months
  Neonatal asphyxia define as fetal death, neonatal death, NICU transfer, neonatal seizure, umbilical-artery blood pH ≤ 7.05 with a base deficit ≥ 12 mmol per liter, intubation for ventilation at delivery or neonatal encephalopathy

CONTACTS AND LOCATIONS:
Overall Officials: Muriel DORET, Pr, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Department of obstetrics, Femme Mère Enfant Hospital, Lyon, France